CLINICAL TRIAL: NCT04701918
Title: A Multicenter, Single-Arm Open Label Phase II Trial of Cryoablation in Combination With Pembrolizumab or Avelumab in Patients With Metastatic Urothelial Carcinoma
Brief Title: Cryoablation With Pembrolizumab Or Avelumab In Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Principal Investigator, Eric Wehrenberg-Klee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-531
Record Dates: First submitted 2020-12-14; First posted 2021-01-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Urothelial Carcinoma; Bladder Cancer
Keywords: Metastatic Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — pembrolizumab; Cryosurgery; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab/Avelumab + Cryoablation (Experimental): If patient is receiving pembrolizumab: Participants will be given 200 mg pembrolizumab intravenously once every 3 weeks. This will continue for up to 2 years as per standard of care. Participants will receive cryoablation between the 1st and 2nd doses of pembrolizumab. Cryoablation consists of using a CT scan to guide one or more thin needles to the tumor through your skin, where extreme cold is applied.
  If patient is receiving avelumab: Participants will be given 800 mg avelumab intravenously once every 2 weeks. This will continue for up to 2 years as per standard of care. Participants will receive cryoablation between the 1st and 2nd doses of avelumab. Cryoablation consists of using a CT scan to guide one or more thin needles to the tumor through your skin, where extreme cold is applied.
  Interventions: Drug: Pembrolizumab; Procedure: Cryoablation; Drug: Avelumab

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous injection through a vein (IV) every 3 weeks
  Other Names: Keytruda
Procedure: Cryoablation — Needle inserted through the skin and into the tumor using CT guidance
Drug: Avelumab — Intravenous injection through a vein (IV) every 2 weeks
  Other Names: Bavencio

SUMMARY:
This research study is examining the effectiveness of pembrolizumab plus cryoablation or aveluma plus cryoablation on people with urothelial carcinoma, including bladder cancer, that has spread.

DETAILED DESCRIPTION:
This is an open label Phase 2, single-arm, multi-institutional clinical trial designed to study the combination of pembrolizumab and cryoablation or avelumab and cryoablation on people with urothelial carcinoma, including bladder cancer, that has spread.

The U.S. Food and Drug Administration (FDA) has approved both cryoablation, pembrolizumab, and avelumab as treatment options for urothelial carcinoma, including bladder cancer, that has spread. However, the FDA has not yet approved the combination of the drugs, pembrolizumab or avelumab, and intervention, cryoablation, for urothelial carcinoma, including bladder cancer, that has spread.

Pembrolizumab is believed to work by binding to a chemical called PD-1 that is found on a special type of white blood cell in your body. Avelumab is believed to work by binding a similar molecule called PD-L1. This may help your body to be better at finding and destroying tumor cells.

Cryoablation is an intervention which may kill cancer cells using extreme cold. It may help the immune system better recognize tumors and act against it.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

Participants will receive study treatment as long as their disease does not get worse or they do not have any unacceptable side effects for up to two years. Participants will be followed for up to 2 years after ending the study treatment.

It is expected that about 30 people will take part in this research study.

Biocompatibles UK Ltd, a device company under Boston Scientific, is supporting this research study by providing funding for the needles used in the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* The subject has read, signed and dated the Informed Consent Form (ICF), having been advised of the risks and benefits of the trial in a language understood by the subject.
* Age > 18 years at date of ICF signature having the ability to comply with the protocol.
* Proof of medical insurance coverage.
* Histologically or cytologically documented metastatic (M1, Stage IV) urothelial carcinoma (including renal pelvis, ureters, urinary bladder, urethra)
* Measurable metastatic disease with at least one site of metastatic disease > 2 cm in size and amenable to percutaneous image-guided cryoablation based on routine Interventional Radiology criteria. Metastasis sites amenable to cryoablation to include lymph node, peritoneum, liver, soft tissue, adrenal glands, kidney, lung, and bone. Must have measurable disease (by RECIST v1.1) independent of the lesion to be ablated (ie patient must have more than one metastasis)
* Life expectancy > 12 weeks.
* PS ECOG 0 or 1
* Laboratory requirements:

  * ANC > 1 x 109/L
  * Platelets > 75 x 109/L
  * ALT / AST < 5 x ULN
  * Total bilirubin <3 mg/dL
  * INR <1.7
  * CrCl >30 ml/min

Exclusion Criteria:

* Lesion to undergo cryoablation cannot have had prior radiation therapy or other locoregional therapy
* Inability to lie flat for the cryoablation procedure.
* Known significant immunodeficiency due to underlying illness (e.g. HIV / AIDS) and/or blood CD4+ T cells <200/ul
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjogren's syndrome, Guillain- Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this trial.
* Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this trial.
* Patients with history of vitiligo and controlled psoriasis are eligible for the trial.
* Continued adverse events from a previously administered chemotherapeutic agents.

Grade 1 adverse events and ongoing toxicities such as alopecia are exempt

* Treatment with systemic corticosteroids exceeding the equivalent of 10 mg/day of prednisone or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial
* Patients who receive acute, low-dose, systemic corticosteroid medications (e.g., a onetime dose of dexamethasone for nausea) or for prevention of hypersensitivity reactions to contrast agents may be enrolled in the trial.
* Anticoagulant or anti-platelet medication that cannot be interrupted prior to cryoablation
* Pregnant or lactating
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or that could affect the interpretation of the results or render the patient at high risk from treatment complications.
* Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including but not limited to IFNs, interleukin [IL]-2) within 6 weeks or five half- lives of the drug, whichever was shorter, prior to Day 1.
* Signs or symptoms clinically significant of infection within 2 weeks prior to Day 1.
* Any other systemic anti-cancer treatment (including investigational agents) within 4 weeks prior to the first dose of study drug. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | up to 2 years
  Evaluate objective response rate of non-ablated lesion(s) for combination pembrolizumab/avelumab and adjunctive cryoablation per RECIST v1.1 criteria

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | up to 2 years
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.
Progression-Free Survival (PFS) | up to 2 years
  Defined using RECIST v1.1
Overall survival (OS) | up to 2 years
  Reported with Kaplan Meier estimates.
Duration of response (DOR) | up to 2 years
  Defined using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wehrenberg-Klee, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation